CLINICAL TRIAL: NCT03283189
Title: Perception of the Risk Associated With the Use of Cosmetics Products During Pregnancy - a Qualitative Study
Brief Title: Cosmetics and Pregnancy
Acronym: PERICOS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Agence Régionale de Santé Rhône-Alpes (Other); Université d'Auvergne (Other); Observatoire Régional de Santé Auvergne-Rhône Alpes (ORS- ARA) (Unknown)
Responsible Party: Sponsor
Other Study IDs: CHU-350
Record Dates: First submitted 2017-09-08; First posted 2017-09-14 (Actual); Last update posted 2019-02-04 (Actual); Status verified 2019-02

CONDITIONS: Pregnancy
Keywords: Use of cosmetics; Pregnant women; Risk perception; Preventive attitude; Qualitative study

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Group 1: Pregnancy follow-up in the only maternity type III of the region (CHU) and in an urban area (around Clermont-Ferrand)
  Interventions: Other: Group discussions
- Group 2: Pregnancy follow-up in the only maternity type III of the region (CHU) and in an urban area (around Clermont-Ferrand)
  Interventions: Other: Group discussions
- Group 3: Pregnancy follow-up in the only private maternity (type II) of the region and in an urban area (around Clermont-Ferrand)
  Interventions: Other: Group discussions
- Group 4: Pregnancy follow-up in the only private maternity (type II) of the region and in an urban area (around Clermont-Ferrand)
  Interventions: Other: Group discussions
- Group 5: Pregnancy follow-up in a type I maternity and in a rural area (around Saint-Flour)
  Interventions: Other: Group discussions
- Group 6: Liberal follow-up of pregnancy

INTERVENTIONS:
Other: Group discussions — The focus group discussions will be conducted in a private room in the maternity of the women. They will last approximately 2 hours and will be led by an interviewer using an interview grid. All interviews will be audio-recorded.
  Groups: Group 1; Group 2; Group 3; Group 4; Group 5

SUMMARY:
The use of cosmetics is an important source of exposure to many chemicals including endocrine disruptors. Recently, national and international scientific recommendations have been issued to limit exposure to chemicals during pregnancy. However, the perception and the use of cosmetics by pregnant women is still little studied. The objectives of the PERICOS study are to identify the risk perception and the attitudes regarding cosmetic's use by the pregnant women.

Understanding the risk perception, the knowledge, attitudes and expectations of women about the use of cosmetics during pregnancy will help to set up effective strategies to improve prevention of chemical exposure.

DETAILED DESCRIPTION:
A qualitative study of 60 pregnant women using six focus groups (9-11 pregnant women per group) was implemented study in Auvergne Region, France. Six focus groups will be conducted until data saturation.

The women will be recruited from the Clermont-Ferrand University Hospital (maternity type III - 2 groups), the private clinic in Beaumont (maternity type II - 2 groups), the Saint-Flour hospital center (maternity type I - 1 group), and from liberal health professionals (1 group).

If a women is found to be eligible, she will be invited to participate in the study. The focus group discussions will be conducted in a private room in the maternity of the women. They will last approximately 2 hours and will be led by an interviewer using an interview grid.

All interviews will be audio-recorded, transcribed, coded and computerized for analysis with the NVIVO v11 software.

ELIGIBILITY:
Inclusion Criteria:

* - Pregnant women between 22 (≥ 22 weeks) et ≤ 39 weeks of gestation;
* Obstetric management in the Réseau de Santé en Périnatalité d'Auvergne (RSPA);
* At least 18 years;
* Understanding and speaking French;
* And giving their signed agreement of participation.

Exclusion Criteria:

* Refusal to participate or to be registered during the collective interview;
* Women with fetal death in utero or whose fetus or fetuses have a malformation;
* Women with psychiatric disorders, mental confusion or language disorders making impossible the interview;
* Women with chronic dermatological pathology requiring dermatological care (eczema, psoriasis, etc.).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: pregnant women
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2019-02-28 (Estimated); Primary Completion 2019-12-30 (Estimated); Study Completion 2019-12-30 (Estimated)

PRIMARY OUTCOMES:
Pregnant women's views on the risk related to the use of cosmetics | at day 1 (during the interview)
  the perception of the risks linked to the use of cosmetics in general, and creams for striae gravidarum in particular, were investigated during the focus groups interviews.

SECONDARY OUTCOMES:
Cosmetic's use during pregnancy | at day 1 (during the interview)
  How cosmetics (all cosmetics and creams for striae gravidarum) are used and modifications in the behavior of pregnant women (decrease of use, choice of other products, etc.). Investigated during the focus groups with a semi-structured interview. All information will be gathered at the time of the interview.
Expectations of pregnant women in terms of information about the use of cosmetics | at day 1 (during the interview)
  needs and expectations of pregnant women in terms of information support and advice about the use of cosmetics were investigated during the focus groups with a semi-structured interview. All information will be gathered at the time of the interview

CONTACTS AND LOCATIONS:
Overall Officials: Cécile MARIE, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France